CLINICAL TRIAL: NCT00005274
Title: Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection (P2C2)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1301
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2005-10

CONDITIONS: Acquired Immunodeficiency Syndrome; Lung Diseases; Cardiovascular Diseases; Heart Diseases; Heart Failure; HIV Infections; Cytomegalovirus Infections; Pneumocystis Carinii Infections; Ebstein-Barr Virus Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Lung Diseases; Cardiovascular Diseases; Heart Diseases; Heart Failure; HIV Infections; Cytomegalovirus Infections; Pneumocystis Infections

SUMMARY:
To determine the prevalence and natural history of pulmonary and cardiac complications associated with HIV infection in utero, in infancy, and during early childhood.

DETAILED DESCRIPTION:
BACKGROUND:

In 1982, a year after the discovery of AIDS in adults, cases were described in children. Subsequent reports clearly indicated that pulmonary and cardiac diseases contributed significantly to morbidity and mortality in children infected with the human immunodeficiency virus.

The initiative was developed by the staff of the Division of Lung Diseases and the Division of Heart and Vascular Diseases after consultation with members of the pulmonary, cardiology, and pediatric communities. The Request for Proposals was released in August 1988 and awards made in May 1989.

DESIGN NARRATIVE:

In this prospective natural history study, research was conducted on the response of the immature lung to Pneumocystis carinii and other opportunistic lung infections, as well as on the etiology and pathogenesis of lymphocytic pulmonary disorders. The types, incidence, course, outcome, and origin of cardiac disorders were also determined. In addition to the pulmonary and cardiovascular measurements, data on the effects of co-infection with other viruses, CMV and EBV, were obtained.

Enrollment of participants began in May 1990 and continued through April 1993 in Group I and through January 1994 for Group II. The cohort was followed at specified intervals for an additional three years beyond the end of recruitment for clinical examination, cardiac, pulmonary, immunologic, and infectious studies and for intercurrent illnesses (The cohorts were followed through January 1997). Follow-up ranged from 2.5 to 6.6 years. The study ends in July 2002. Analysis of the database, preparation of manuscripts and follow-up of adult type pulmonary function studies in infants currently followed at sites conducting the Womens & Infants Transmission Study (WITS) continue through July 2002

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-05; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kaplan — University of California; Meyer Kattan — Icahn School of Medicine at Mount Sinai; D. Kutner — The Cleveland Clinic; Stephen Lipschultz — Children's Hospital Medical Center, Cincinnati; Robert Mellins — Presbyterian Hospital; William Shearer — Baylor College of Medicine; David Teitel — University of California

REFERENCES:
- [Background] Shearer WT, Rosenblatt HM, Schluchter MD, Mofenson LM, Denny TN. Immunologic targets of HIV infection: T cells. NICHD IVIG Clinical Trial Group, and the NHLBI P2C2 Pediatric Pulmonary and Cardiac Complications of HIV Infection Study Group. Ann N Y Acad Sci. 1993 Oct 29;693:35-51. doi: 10.1111/j.1749-6632.1993.tb26255.x. PMID 7903519
- [Background] Cohen HL, Davis L, Hunter J, Carp D, Geromanos K, Sunkle S. Coordinating a large multicentered HIV research project. J Assoc Nurses AIDS Care. 1997 Jan-Feb;8(1):41-50. doi: 10.1016/S1055-3290(97)80036-2. PMID 9085248
- [Background] The P2C2 HIV Study Group. The pediatric pulmonary and cardiovascular complications of vertically transmitted human immunodeficiency virus (P2C2 HIV) infection study: design and methods. The P2C2 HIV Study Group. J Clin Epidemiol. 1996 Nov;49(11):1285-94. doi: 10.1016/s0895-4356(96)00230-2. PMID 8892497
- [Background] Pitt J, Goldfarb J, Schluchter M, Kovacs A, Cooper E, Hodes D, McIntosh K, Peavy H, Shearer W. HIV vertical transmission rate determinations are subject to differing definitions and therefore different rates. The Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection Study Group. J Clin Epidemiol. 1998 Feb;51(2):159-64. doi: 10.1016/s0895-4356(97)00239-4. PMID 9474076
- [Background] Martin R, Boyer P, Hammill H, Peavy H, Platzker A, Settlage R, Shah A, Sperling R, Tuomala R, Wu M. Incidence of premature birth and neonatal respiratory disease in infants of HIV-positive mothers. The Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted Human Immunodeficiency Virus Infection Study Group. J Pediatr. 1997 Dec;131(6):851-6. doi: 10.1016/s0022-3476(97)70032-5. PMID 9427889
- [Background] Shearer WT, Lipshultz SE, Easley KA, McIntosh K, Pitt J, Quinn TC, Kattan M, Goldfarb J, Cooper E, Bryson Y, Kovacs A, Bricker JT, Peavy H, Mellins RB, Heart N, Institute LB. Alterations in cardiac and pulmonary function in pediatric rapid human immunodeficiency virus type 1 disease progressors. Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted Human Immunodeficiency Virus Study Group. Pediatrics. 2000 Jan;105(1):e9. doi: 10.1542/peds.105.1.e9. PMID 10617746
- [Background] Kovacs A, Schluchter M, Easley K, Demmler G, Shearer W, La Russa P, Pitt J, Cooper E, Goldfarb J, Hodes D, Kattan M, McIntosh K. Cytomegalovirus infection and HIV-1 disease progression in infants born to HIV-1-infected women. Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection Study Group. N Engl J Med. 1999 Jul 8;341(2):77-84. doi: 10.1056/NEJM199907083410203. PMID 10395631
- [Background] Starc TJ, Langston C, Goldfarb J, Colin AA, Cooper ER, Easley KA, Sunkle S, Schluchter MD. Unexpected non-HIV causes of death in children born to HIV-infected mothers. Pediatric Pulmonary and Cardiac Complications of Vertically Transmitted HIV Infection Study Group. Pediatrics. 1999 Jul;104(1):e6. doi: 10.1542/peds.104.1.e6. PMID 10390292
- [Background] Jenson H, McIntosh K, Pitt J, Husak S, Tan M, Bryson Y, Easley K, Shearer W. Natural history of primary Epstein-Barr virus infection in children of mothers infected with human immunodeficiency virus type 1. J Infect Dis. 1999 Jun;179(6):1395-404. doi: 10.1086/314764. PMID 10228060
- [Background] Lai WW, Lipshultz SE, Easley KA, Starc TJ, Drant SE, Bricker JT, Colan SD, Moodie DS, Sopko G, Kaplan S. Prevalence of congenital cardiovascular malformations in children of human immunodeficiency virus-infected women: the prospective P2C2 HIV Multicenter Study. P2C2 HIV Study Group, National Heart, Lung, and Blood Institute, Bethesda, Maryland. J Am Coll Cardiol. 1998 Nov 15;32(6):1749-55. doi: 10.1016/s0735-1097(98)00449-5. PMID 9822105
- [Background] Cleveland RH, Schluchter M, Wood BP, Berdon WE, Boechat MI, Easley KA, Meziane M, Mellins RB, Norton KI, Singleton E, Trautwein L. Chest radiographic data acquisition and quality assurance in multicenter studies. Pediatr Radiol. 1997 Nov;27(11):880-7. doi: 10.1007/s002470050262. PMID 9361051
- [Background] Starc TJ, Lipshultz SE, Kaplan S, Easley KA, Bricker JT, Colan SD, Lai WW, Gersony WM, Sopko G, Moodie DS, Schluchter MD. Cardiac complications in children with human immunodeficiency virus infection. Pediatric Pulmonary and Cardiac Complications of Vertically Transmitted HIV Infection (P2C2 HIV) Study Group, National Heart, Lung, and Blood Institute. Pediatrics. 1999 Aug;104(2):e14. doi: 10.1542/peds.104.2.e14. PMID 10429132
- [Background] Pitt J, Schluchter M, Jenson H, Kovacs A, LaRussa P, McIntosh K, Boyer P, Cooper E, Goldfarb J, Hammill H, Hodes D, Peavy H, Sperling R, Tuomala R, Shearer W. Maternal and perinatal factors related to maternal-infant transmission of HIV-1 in the P2C2 HIV study: the role of EBV shedding. Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV-1 Infection (P2C2 HIV) Study Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Dec 15;19(5):462-70. doi: 10.1097/00042560-199812150-00004. PMID 9859959
- [Background] Xanthos GJ, Carp D, Geromanos KL. Recognizing nurses' contributions to the clinical research process. J Assoc Nurses AIDS Care. 1998 Jan-Feb;9(1):39-48. doi: 10.1016/S1055-3290(98)80075-7. PMID 9436166
- [Background] Platzker AC, Colin AA, Chen XC, Hiatt P, Hunter J, Koumbourlis AC, Schluchter MD, Ting A, Wohl ME. Thoracoabdominal compression and respiratory system compliance in HIV-infected infants. Am J Respir Crit Care Med. 2000 May;161(5):1567-71. doi: 10.1164/ajrccm.161.5.9902066. PMID 10806156
- [Background] Saidi AS, Moodie DS, Garson A Jr, Lipshultz SE, Kaplan S, Lai WW, Colan SD, Starc TJ, Shanbhag S, Easley KA, Bricker JT. Electrocardiography and 24-hour electrocardiographic ambulatory recording (Holter monitor) studies in children infected with human immunodeficiency virus type 1. The Pediatric Pulmonary and Cardiac Complications of Vertically Transmitted HIV-1 Infection Study Group. Pediatr Cardiol. 2000 May-Jun;21(3):189-96. doi: 10.1007/s002460010038. PMID 10818172
- [Background] Lipshultz SE, Easley KA, Orav EJ, Kaplan S, Starc TJ, Bricker JT, Lai WW, Moodie DS, McIntosh K, Schluchter MD, Colan SD. Left ventricular structure and function in children infected with human immunodeficiency virus: the prospective P2C2 HIV Multicenter Study. Pediatric Pulmonary and Cardiac Complications of Vertically Transmitted HIV Infection (P2C2 HIV) Study Group. Circulation. 1998 Apr 7;97(13):1246-56. doi: 10.1161/01.cir.97.13.1246. PMID 9570194
- [Background] Lipshultz SE, Easley KA, Orav EJ, Kaplan S, Starc TJ, Bricker JT, Lai WW, Moodie DS, Sopko G, McIntosh K, Colan SD. Absence of cardiac toxicity of zidovudine in infants. Pediatric Pulmonary and Cardiac Complications of Vertically Transmitted HIV Infection Study Group. N Engl J Med. 2000 Sep 14;343(11):759-66. doi: 10.1056/NEJM200009143431102. PMID 10984563
- [Background] Langston C, Cooper ER, Goldfarb J, Easley KA, Husak S, Sunkle S, Starc TJ, Colin AA; P2C2 HIV Study Group. Human immunodeficiency virus-related mortality in infants and children: data from the pediatric pulmonary and cardiovascular complications of vertically transmitted HIV (P(2)C(2)) Study. Pediatrics. 2001 Feb;107(2):328-38. doi: 10.1542/peds.107.2.328. PMID 11158466
- [Background] Lipshultz SE, Easley KA, Orav EJ, Kaplan S, Starc TJ, Bricker JT, Lai WW, Moodie DS, Sopko G, Colan SD. Cardiac dysfunction and mortality in HIV-infected children: The Prospective P2C2 HIV Multicenter Study. Pediatric Pulmonary and Cardiac Complications of Vertically Transmitted HIV Infection (P2C2 HIV) Study Group. Circulation. 2000 Sep 26;102(13):1542-8. doi: 10.1161/01.cir.102.13.1542. PMID 11182983
- [Background] Alderson PO, Chen DC, Fleishman MJ, Hoh CK, Kim CK, Lee VW, Mellins RB, Miller JH, Moore WH, Peavy HH, Shah A, Treves ST. Radioaerosol scintigraphy in infants and children born to mothers with HIV disease. Pediatric Pulmonary and Cardiovascular Complications (of Vertically Transmitted Human Immunodeficiency Virus) Study Group. Radiology. 1999 Mar;210(3):815-22. doi: 10.1148/radiology.210.3.r99mr09815. PMID 10207486
- [Background] Hornberger LK, Lipshultz SE, Easley KA, Colan SD, Schwartz M, Kaplan S, Starc TJ, Ayres NA, Lai WW, Moodie DS, Kasten-Sportes C, Sanders SP. Cardiac structure and function in fetuses of mothers infected with HIV: the prospective PCHIV multicenter study. Am Heart J. 2000 Oct;140(4):575-84. doi: 10.1067/mhj.2000.109645. PMID 11011330
- [Background] Lai WW, Colan SD, Easley KA, Lipshultz SE, Starc TJ, Bricker JT, Kaplan S; P2C2 HIV Study Group, National Heart, Lung, and Blood Institute. Dilation of the aortic root in children infected with human immunodeficiency virus type 1: The Prospective P2C2 HIV Multicenter Study. Am Heart J. 2001 Apr;141(4):661-70. doi: 10.1067/mhj.2001.113757. PMID 11275935
- [Background] Demmler GJ, Istas A, Easley KA, Kovacs A. Results of a quality assurance program for detection of cytomegalovirus infection in the pediatric pulmonary and cardiovascular complications of vertically transmitted human immunodeficiency virus infection study. J Clin Microbiol. 2000 Nov;38(11):3942-5. doi: 10.1128/JCM.38.11.3942-3945.2000. PMID 11060049
- [Background] Cohen H, Chen XC, Sunkle S, Davis L, Geromanos K, Xanthos G, Shearer W. Ability of caregivers to read delayed hypersensitivity skin tests in children exposed to and infected by HIV. The Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Study Group. J Pediatr Health Care. 2000 Mar-Apr;14(2):50-5. doi: 10.1067/mph.2000.101341. PMID 10736138
- [Background] Lipshultz SE, Easley KA, Orav EJ, Kaplan S, Starc TJ, Bricker JT, Lai WW, Moodie DS, Sopko G, Schluchter MD, Colan SD. Reliability of multicenter pediatric echocardiographic measurements of left ventricular structure and function: the prospective P(2)C(2) HIV study. Circulation. 2001 Jul 17;104(3):310-6. doi: 10.1161/01.cir.104.3.310. PMID 11457750
- [Background] Meyers A, Shah A, Cleveland RH, Cranley WR, Wood B, Sunkle S, Husak S, Cooper ER. Thymic size on chest radiograph and rapid disease progression in human immunodeficiency virus 1-infected children. Pediatr Infect Dis J. 2001 Dec;20(12):1112-8. doi: 10.1097/00006454-200112000-00004. PMID 11740315
- [Background] Keesler MJ, Fisher SD, Lipshultz SE. Cardiac manifestations of HIV infection in infants and children. Ann N Y Acad Sci. 2001 Nov;946:169-78. doi: 10.1111/j.1749-6632.2001.tb03911.x. PMID 11762985
- [Background] Miller TL, Easley KA, Zhang W, Orav EJ, Bier DM, Luder E, Ting A, Shearer WT, Vargas JH, Lipshultz SE; Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection (P2C2 HIV) Study Group; National Heart, Lung, and Blood Institute, Bethesda, MD. Maternal and infant factors associated with failure to thrive in children with vertically transmitted human immunodeficiency virus-1 infection: the prospective, P2C2 human immunodeficiency virus multicenter study. Pediatrics. 2001 Dec;108(6):1287-96. doi: 10.1542/peds.108.6.1287. PMID 11731650
- [Background] Starc TJ, Lipshultz SE, Easley KA, Kaplan S, Bricker JT, Colan SD, Lai WW, Gersony WM, Sopko G, Moodie DS, Schluchter MD. Incidence of cardiac abnormalities in children with human immunodeficiency virus infection: The prospective P2C2 HIV study. J Pediatr. 2002 Sep;141(3):327-34. doi: 10.1067/mpd.2002.126301. PMID 12219051
- [Background] Jenson HB, Gauntt CJ, Easley KA, Pitt J, Lipshultz SE, McIntosh K, Shearer WT; Pediatric Pulmonary and Cardiovascular Complication of HIV-1 Infection Study Group. Evaluation of coxsackievirus infection in children with human immunodeficiency virus type 1-associated cardiomyopathy. J Infect Dis. 2002 Jun 15;185(12):1798-802. doi: 10.1086/340819. Epub 2002 May 31. PMID 12085328
- [Background] Lipshultz SE, Easley KA, Orav EJ, Kaplan S, Starc TJ, Bricker JT, Lai WW, Moodie DS, Sopko G, Schluchter MD, Colan SD; Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection (P(2)C(2) HIV) Study Group. Cardiovascular status of infants and children of women infected with HIV-1 (P(2)C(2) HIV): a cohort study. Lancet. 2002 Aug 3;360(9330):368-73. doi: 10.1016/S0140-6736(02)09607-1. PMID 12241776
- [Background] Rivenes SM, Colan SD, Easley KA, Kaplan S, Jenkins KJ, Khan MN, Lai WW, Lipshultz SE, Moodie DS, Starc TJ, Sopko G, Zhang W, Bricker JT; Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection Study Group. Usefulness of the pediatric electrocardiogram in detecting left ventricular hypertrophy: results from the Prospective Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection (P2C2 HIV) multicenter study. Am Heart J. 2003 Apr;145(4):716-23. doi: 10.1067/mhj.2003.15. PMID 12679770
- [Background] Colin AA, Sunil Rao J, Chen XC, Hunter JM, Hanrahan J, Hiatt P, Kattan M, Koumbourlis A, Mellins RB, Peavy HH, Platzker A, Ting A, Steinbach S, Wohl ME; Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted Human Immunodeficiency Virus Study Group, National Heart, Lung, and Blood Institute. Forced expiratory flow in uninfected infants and children born to HIV-infected mothers. Am J Respir Crit Care Med. 2001 Mar;163(4):865-73. doi: 10.1164/ajrccm.163.4.9901040. PMID 11282758
- [Background] Kearney DL, Perez-Atayde AR, Easley KA, Bowles NE, Bricker JT, Colan SD, Kaplan S, Lai WW, Lipshultz SE, Moodie DS, Sopko G, Starc TJ, Towbin JA; Pediatric Pulmonary and Cardiovascular Complication of Vertically Transmitted HIV Infected (P2C2 HIV) Study Group, National Heart, Lung and Blood Institute. Postmortem cardiomegaly and echocardiographic measurements of left ventricular size and function in children infected with the human immunodeficiency virus. The Prospective P2C2 HIV Multicenter Study. Cardiovasc Pathol. 2003 May-Jun;12(3):140-8. doi: 10.1016/s1054-8807(03)00035-8. PMID 12763553
- [Background] Perez-Atayde AR, Kearney DI, Bricker JT, Colan SD, Easley KA, Kaplan S, Lai WW, Lipshultz SE, Moodie DS, Sopko G, Starc TJ; P2C2 HIV Study Group. Cardiac, aortic, and pulmonary arteriopathy in HIV-infected children: the Prospective P2C2 HIV Multicenter Study. Pediatr Dev Pathol. 2004 Jan-Feb;7(1):61-70. doi: 10.1007/s10024-003-1001-9. PMID 15255036
- [Background] Fisher SD, Easley KA, Orav EJ, Colan SD, Kaplan S, Starc TJ, Bricker JT, Lai WW, Moodie DS, Sopko G, Lipshultz SE; Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection (P2C2 HIV) Study Group. Mild dilated cardiomyopathy and increased left ventricular mass predict mortality: the prospective P2C2 HIV Multicenter Study. Am Heart J. 2005 Sep;150(3):439-47. doi: 10.1016/j.ahj.2005.06.012. PMID 16169321
- [Background] Geromanos K, Sunkle SN, Mauer MB, Carp D, Ancker J, Zhang W, Easley KA, Schluchter MD, Kozinetz CA, Mellins RB. Successful techniques for retaining a cohort of infants and children born to HIV-infected women: the prospective P2C2 HIV study. J Assoc Nurses AIDS Care. 2004 Jul-Aug;15(4):48-57. doi: 10.1177/1055329003256653. PMID 15296658
- Available data/document: Individual Participant Data Set: P2C2 — http://biolincc.nhlbi.nih.gov/studies/p2c2/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/p2c2/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/p2c2/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/p2c2/